CLINICAL TRIAL: NCT04402073
Title: Personalized Risk-Adapted Therapy in Post-Pubertal Patients With Newly-Diagnosed Medulloblastoma (PersoMed-I)
Brief Title: Personalized Risk-Adapted Therapy in Post-Pubertal Patients With Newly-Diagnosed Medulloblastoma
Acronym: PersoMed-I
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1634
Record Dates: First submitted 2020-04-01; First posted 2020-05-26 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Medulloblastoma
Keywords: brain; medullobalstoma; MRI; radiotherapy; biomarkers
MeSH Terms: conditions — Medulloblastoma | interventions — sonidegib; Cisplatin; Lomustine; Vincristine; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Phase II, comparative, randomized (experimental : standard arm 1:1, no blinding, no active or placebo control, parallel group, therapeutic
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- standard arms (Other): Criteria: Adult SHH (p53wt) M0-1, adult WNT M0-1, adult Group 4 M0-1.
  Radiotherapy to the cranio-spinal axis of 35.2 Gy in 22 daily fractions of 1.6 Gy, followed by an additional boost to the tumour site of 19.8 Gy in 11 daily fractions of 1.8 Gy, summing up to a total dose of 55.0 Gy in 33 daily fractions of 1.6/1.8 Gy.
  Criteria: Post pubertal < 18 y SHH (p53wt) M0.
  Radiotherapy to the cranio-spinal axis of 23.4 Gy in 13 daily fractions of 1.8 Gy, followed by an additional boost to the tumour site of 30.6 Gy in 17 daily fractions of 1.8 Gy, summing up to a total dose of 54.0 Gy in 30 daily fractions of 1.8 Gy.
  Interventions: Drug: Cisplatin; Drug: Lomustine; Drug: Vincristine; Radiation: radiotherapy
- experimental arms (Experimental): Radiotherapy Criteria: Adult and post-pubertal SHH (p53wt) M0; adult WNT M0, adult Group 4 M0.
  Radiotherapy to the cranio-spinal axis of 23.4 Gy in 13 daily fractions of 1.8 Gy, followed by an additional boost to the tumour site of 30.6 Gy in 17 daily fractions of 1.8 Gy, summing up to a total dose of 54.0 Gy in 30 daily fractions of 1.8 Gy.
  SMO-inhibitor Criteria: Adult and post-pubertal SHH (p53wt) M0.
  Sonidegib 200 mg/day (daily) from first day of radio-chemotherapy until end of maintenance chemotherapy, including 6w chemotherapy break.
  Interventions: Drug: Sonidegib; Drug: Cisplatin; Drug: Lomustine; Drug: Vincristine; Radiation: radiotherapy

INTERVENTIONS:
Drug: Sonidegib — Sonidegib is a selective smoothened inhibitor that inhibits the sonic hedgehog-signaling pathway. It is used in patients with locally advanced basal cell carcinoma (BCC) that has recurred following surgery or radiation therapy, or those who are not candidates for surgery or radiation therapy.
  Arms: experimental arms
Drug: Cisplatin — Cisplatin (CIS) is a platinum derivate used in the treatment in several epithelial tumours. The application route is through the veins.
Drug: Lomustine — Lomustine is a nitrosourea used in the treatment of brain tumours and Hodgkin's disease. The application route is oral.
Drug: Vincristine — Vincristine sulfate (VCR) is an inhibitor of microtubule formation in the mitotic spindle, resulting in an arrest of dividing cells at the metaphase stage. Vincristine sulfate is indicated in acute leukemia, Hodgkin's disease, non-Hodgkin's lymphomas, rhabdomyosarcoma, neuroblastoma, and Wilms' tumor. The application route is through the vein.
Radiation: radiotherapy — Radiotherapy to the cranio-spinal axis of 35.2 Gy in 22 daily fractions of 1.6 Gy, followed by an additional boost to the tumour site of 19.8 Gy in 11 daily fractions of 1.8 Gy, summing up to a total dose of 55.0 Gy in 33 daily fractions of 1.6/1.8 Gy.

SUMMARY:
Medulloblastoma is a rare brain malignancy, mainly affecting children. Treatment of this rapidly growing tumor begins with maximal surgical removal plus radiation and chemotherapy. Treatment toxicity is high. Post-pubertal and pediatric medulloblastomas are biologically and prognostically different, which mandates age-adapted treatment strategies. Patients after puberty bear an intermediate to high prognostic risk. This means that a large number of these patients, are faced with death and/or disability (mainly neurocognitive). Therefore, the scientific and medical need is high. One of the genetic subgroups of medulloblastoma, the SHH-subgroup (Sonic HedgeHog- subgroup), is highly overrepresented in medulloblastoma patients after puberty. This subgroup can be treated with a targeted therapy. The investigators will therefore randomize patients and treat SHH-subgroup patients with sonidegib and a reduction of radiotherapy dose in the experimental arm of the trial. The hypothesis that this personalized risk-adapted therapy will improve outcomes in view of increased efficacy and decreased toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, histologically proven, genetically classified, centrally confirmed medulloblastoma (WNT M0-1, SHH M0-1 (p53wt), Group 4 M0-1)
* Molecular subtype: medulloblastoma, SHH-activated and TP53-wildtype, M0-1; medulloblastoma, WNT-activated, M0-1; medulloblastoma, Group 4, M0-1
* Histologic subtype: medulloblastoma, classic (CMB); medulloblastoma, desmoplastic/nodular (DNMB); medulloblastoma, with extensive nodularity (MBEN); medulloblastoma, large cell/anaplastic (LCA)
* Adult (18 years and above): in WNT-activated and Group 4 medulloblastoma
* Post-pubertal, defined as females with a bone age of at least 15 years and males with a bone age of at least 17 years, or adult (greater than 18 y of age) (see appendix N) in SHH-activated and TP53-wildtype medulloblastoma
* Availability of prognostic markers (MYC/MYCN amplification, MYC/MYCN mutation)
* Availability of paraffin embedded tumour tissue (FFPE) (1 block or 30 unstained slides) and whole blood sample (10 ml) for central review
* For patients with SHH activated tumours: exclusion of germline alteration of TP53, PTCH, SUFU, BRCA2 and PALB2 if known before randomization
* Clinical status within 2 weeks of randomization: Karnofsky 50-100. NANO-score 0 to 9 (allowing full-blown cerebellar symptoms)
* Clinically standard-risk (centrally assessed MRI review) defined as: total or near total surgical resection with less than or equal to 1.5 cm2 (measured in axial plane) of residual tumour on early post-operative MRI, without and with contrast; no CNS metastasis on MRI (cranial and spinal); Chang stage M0-1 with no clinical evidence of extra-CNS metastasis
* Full recovery from surgery or any post-surgical complication (e.g. Bleeding, infections etc)
* Pre-surgery and/or post-surgery MRI available.
* Baseline brain MRI and spinal MRI available within 2 weeks of randomization.
* Normal liver, renal and haematological function within 2 weeks of randomization.
* WBC greater than or equal to 3×10^9/L
* ANC greater than or equal to 1.5×10^9/L
* Platelet count of greater than or equal to 100×10^9/L independent of transfusion
* Hemoglobin greater than or equal to 10 g/dl
* Total Bilirubin less than or equal to 1.5 ULN
* ALT (SGPT), AST (SGOT), alkaline phosphatase (ALP) less than or equal to 2.5 × ULN
* Serum creatinine less than 1.5 x ULN or creatinine clearance (CrCl) greater than 30 mL/min (using the Cockcroft-Gault formula)
* Negative serum or urine pregnancy test within 7 days of randomization for WOCBP.
* Patients of childbearing / reproductive potential (WOCBP) must use two methods of adequate birth control, including a highly effective method and a barrier method during the study treatment period and for at least 20 months after the last study treatment is mandatory for the patients that received sonidegib, for all other patients this period is at least 6 months after the last study treatment. A highly effective method of birth control is defined as those which result in low failure rate (i.e. less than 1% per year) when used consistently and correctly. Male patients even those who have had a vasectomy must always use a condom during treatment and for 6 months after last treatment. Men should not donate semen during treatment and for at least 6 months after ending treatment (donation of semen for the semen analyses of the fertility project 1 b is allowed). Appendix H.
* Female subjects who are breast feeding must discontinue nursing prior to the first dose of study treatment and until 20 months after the last study treatment.
* Before patient registration/randomization, written informed consent must be given according to ICH/GCP, and national/local regulations. For patients less than 18 years of age, consent has to be obtained from the parent(s) or legal representative.

Exclusion Criteria:

* Prior treatment for medulloblastoma
* Unavailability of central review pathology results.
* Inability to start radiotherapy within 43 days of surgery
* Significant sensorineural hearing deficit as defined by pure tone audiometry with bone conduction or air conduction and normal tympanogram showing impairment greater than or equal to 20 dB at 1-3 kHz
* Any medical contraindication to radiotherapy or chemotherapy.
* Hypersensitivity to contrast medium for MRI.
* Hypersensitivity towards the active substance of any of study drugs or their excipients
* Prior or current use of mitoxantrone, methotrexate, topotecan, imatinib, irinotecan or statins
* Concurrent severe or uncontrolled medical disease (e.g., active systemic infection, diabetes, psychiatric disorder) that, in the opinion of the investigator, would compromise the safety of the patient or compromise the ability of the patient to complete the study
* Prior or second invasive malignancy, except non-melanoma skin cancer, completely resected cervical carcinoma in situ, low risk prostate cancer (cT1-2a N0 and Gleason score less than or equal to 6 and PSA less than 10 ng/mL), either totally resected or irradiated with curative intent (with PSA of less than or equal to 0.1 ng/mL) or under active surveillance as per ESMO guidelines. Other cancers for which the subject has completed potentially curative treatment more than 5 years prior to diagnosis of medulloblastoma study entry are allowed
* Known history or current evidence of active Hepatitis B (e.g., positive HBV surface antigen) or C (e.g., HCV RNA [qualitative] is detected)
* Known or current evidence of Human Immunodeficiency Virus (HIV) infection (positive HIV-1/2 antibodies)
* Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 91 months after the date of recruitment of the first patient
  compare progression-free survival (PFS) by central review of a personalized intensity-modulated therapy (experimental arm; sonidegib) vs. standard therapy in the SHH-activated subgroup in post-pubertal patients with newly diagnosed standard risk medulloblastoma.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | when 43 PFS events are observed which is estimated to occur 91 months after the date of recruitment of the first patient.
overall survival (OV) | when 43 PFS events are observed which is estimated to occur 91 months after the date of recruitment of the first patient.
safety and tolerability profile: CTCAE | when 43 PFS events are observed which is estimated to occur 91 months after the date of recruitment of the first patient.
  This study will use the International Common Terminology Criteria for Adverse Events (CTCAE), version 5.0, for adverse event reporting (with neurological, kidney, auditory, endocrine and radiotherapy associated as AE of special interest). The highest CTCAE v. 5 grading per cycle and per patient will be computed at the EORTC HQ for analysis . Safety and tolerability analyses will be performed in the safety population. Severe grades (3/4) which did not resolve after treatment discontinuation or emerged during follow-up will be identified and listed.
health-related quality of life (HRQoL) | when 43 PFS events are observed which is estimated to occur 91 months after the date of recruitment of the first patient.
  The primary HRQoL endpoint that is considered relevant for this study is social functioning. The other scales from the QLQ-C30 and BN20 will be considered as exploratory in nature.
  A difference of 10 points on the 100-point QLQ-C30 social functioning scale between the two arms will be considered as clinically relevant.
overall survival | when 43 PFS events are observed which is estimated to occur 91 months after the date of recruitment of the first patient.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hau, Principal Investigator — EORTC study coordinator
Locations (50):
- Australia (10):
  - Royal Adelaide Hospital, Adelaide
  - Princess Alexandra Hospital - University Of Queensland, Brisbane
  - Austin Health - Austin hospital, Melbourne
  - Peter Maccallum Cancer Institute, Melbourne
  - Sir Charles Gairdner Hospital, Nedlands
  - John Hunter Children's Hospital, New Lambton Heights
  - Prince Of Wales Hospital, Sydney
  - Royal North Shore Hospital, Sydney
  - Sydney Children's Hospital, Sydney
  - Westmead Hospital - Crown Princess Mary Cancer Center, Westmead
- Austria (2):
  - A.O Landeskrankenhaus - Innsbruck Universitaetsklinik, Innsbruck
  - AKH unikliniken, Vienna
- France (7):
  - CHRU de Lille, Lille
  - Centre Leon Berard, Lyon
  - Hopital de La Timone (APHM), Marseille
  - CHU de Nice - Hopital Pasteur, Nice
  - Hopital la Pitie-Salpetriere, Paris
  - Institut de Cancerologie de l'Ouest (ICO) - Saint Herblain, Saint-Herblain
  - CHU de Toulouse - Institut Claudius Regaud - IUCT oncopole, Toulouse
- Germany (17):
  - Knappschaft Krankenhaus Langendreer, Bochum
  - Universitaetsklinikum Bonn, Bonn
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - HELIOS Kliniken - HELIOS Klinikum Erfurt GmbH, Erfurt
  - Universitaetsklinikum - Essen, Essen
  - University Frankfurt - Goethe Univ. - University Hospital Frankfurt -Senckenberg Institute of Neurooncology, Frankfurt
  - Universitaetsklinikum Freiburg - Klinik fuer Neurochirurgie, Freiburg im Breisgau
  - Universitaetsmedizin Goettingen - Georg-August Universitaet, Goettigen
  - Universitaets Krankenhaus Eppendorf - Universitaetsklinikum Hamburg-Eppendorf KE - University Cancer Center, Hamburg
  - Universitaetsklinikum Heidelberg - UniversitaetsKlinikum Heidelberg - Head Hospital, Heidelberg
  - Universitaetsklinikum Leipzig-Klinik fuer Strahlentherapie und Radioonkologie, Leipzig
  - Univ. Mainz - Universitaetsmedizin der Johannes Gutenberg Universitaet Mainz-University Medical Center, Mainz
  - UniversitaetsMedizin Mannheim, Mannheim
  - Klinikum Rechts der isar Der Technische Universitaet Muenchen, Munich
  - Ludwig-Maximilians-Universitaet Muenchen - Campus Grosshadern, Munich
  - Universitaetskliniken Regensburg - Universitaetsklinikum Regensburg, Regensburg
  - Universitaetsklinikum Tuebingen- Crona Kliniken, Tübingen
- Italy (5):
  - AUSL Bologna - Ospedale Bellaria, Bologna
  - Univ. of Florence -Azienda Ospedaliero-Universitaria Careggi, Florence
  - IRCCS - Istituto Neurologico Carlo Besta, Milan
  - Azienda Ospedaliera Citta della Salute e della Scienza di Torino, Torino
  - ULSS2 - Marca Trevigniana, Treviso
- Netherlands (2):
  - Universitair Medisch Centrum Groningen, Groningen
  - Erasmus MC, Rotterdam
- Spain (5):
  - Institut Catala d'Oncologia - ICO Badalona - Hospital Germans Trias i Pujol, Badalona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario 12 De Octubre, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois - Lausanne, Lausanne
  - University Hospital zurich, Zurich